CLINICAL TRIAL: NCT03041779
Title: A Single Blinded, Open-labelled, Randomized Control Trial Comparing Acetaminophen Rectal Suppository With Diclofenac Rectal Suppository as Analgesia for Perineal Injury Following Childbirth
Brief Title: Comparison Between Rectal Suppository Acetaminophen and Diclofenac Sodium as Analgesia for Postpartum Perineal Tear
Acronym: SuPPerP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinical Research Centre, Malaysia (Other)
Responsible Party: Principal Investigator, Woon Shu Yuan, Doctor, Clinical Research Centre, Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMRR-15-868-26140
Record Dates: First submitted 2016-12-12; First posted 2017-02-03 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Perineal Tear; Perineal Laceration (Obstetric)
MeSH Terms: interventions — Diclofenac; Suppositories; Acetaminophen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paracetamol (Active Comparator): Paracetamol 500Mg Suppository
  Interventions: Drug: Diclofenac Sodium 50Mg Suppository
- Voltaren (Active Comparator): Diclofenac Sodium 50Mg Suppository
  Interventions: Drug: Paracetamol 500Mg Suppository

INTERVENTIONS:
Drug: Diclofenac Sodium 50Mg Suppository
  Other Names: Voltaren 50Mg Suppository
  Arms: Paracetamol
Drug: Paracetamol 500Mg Suppository
  Other Names: Acetaminophen 500Mg Suppository
  Arms: Voltaren

SUMMARY:
To assess the prevalence of pain score for perineum pain following childbirth followed by phase 2 study to assess the analgesic effectiveness of acetaminophen and diclofenac rectal suppository in postpartum perineum pain secondary to perineal trauma.

DETAILED DESCRIPTION:
Studies has demonstrated that non-steroidal anti-inflammatory drugs (NSAIDs) rectal suppositories are associated with less pain up to 24 hours after birth, and less additional analgesia is required. Therefore, In view of rectal route of analgesic administration is better in local action and systemic paracetamol also proven to be effective in controlling post-partum perineal pain with unknown effectiveness in its suppository form; the investigators would like to conduct this study to investigate the effectiveness of acetaminophen rectal suppository versus diclofenac rectal suppository in controlling postpartum perineal pain. This study will be conducted in 2 stages. Stage 1 is a 3 months prospective observational study which aims to determine the prevalence and severity of perineal pain following childbirth in Hospital Sultanah Aminah, Johor Bahru; while Stage 2 is a single blinded, open-labelled, randomized control trial study design which will determine if acetaminophen rectal suppository is as equivalence as diclofenac rectal suppository in reducing postpartum perineal pain secondary to perineal trauma.

ELIGIBILITY:
Inclusion Criteria:

Stage 1:

a) All pregnant women who sustained perineal trauma (either 1st degree tear, 2nd degree tear or episiotomy) post vaginal delivery

Stage 2:

1. All pregnant women who have planned vaginal delivery in HSAJB from 1st January 2016 till 30th June 2016.
2. All pregnant women who sustained 1st degree/ 2nd degree perineal tear or episiotomy tear post vaginal delivery.
3. All pregnant women who have consented to involve in the study.

Exclusion Criteria:

Stage 1:

1. Patient who sustained additional perineal tear (eg. Labial tear or periurethral tear) following childbirth.
2. Patient who developed post-partum complications.

Stage 2:

1. Patient who is allergic to paracetamol or voltaren.
2. Patient who is unable to or unwilling to give consent.
3. Patient who is ended up with caesarean section.
4. Patient who sustained additional perineal tear including labial tear or periurethral tear.
5. Patient who developed postpartum complications (eg. Retained placenta, uterine atony, postpartum haemorrhage, multiple vaginal wall tear etc. )

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 909 (Actual)
Dates: Start 2015-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
perineum pain score following childbirth | at 2nd to 3rd hour post repair

SECONDARY OUTCOMES:
perineum pain score following childbirth | immediate after delivery
perineum pain score following childbirth | immediate post perineum repair
perineum pain score following childbirth | at 5th to 6th hour post repair
perineum pain score following childbirth | prior to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Shu Yuan Woon, MBBS, Principal Investigator — O&G department, Hospital Sultanah Aminah Johor Bahru, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Cunningham G, Leveno K, Bloom S, et al. Maternal Anatomy. Williams obstetrics. 22nd Edition. New York: McGraw-Hill, 2005:21.
- [Result] Albers L, Garcia J, Renfrew M, McCandlish R, Elbourne D. Distribution of genital tract trauma in childbirth and related postnatal pain. Birth. 1999 Mar;26(1):11-7. doi: 10.1046/j.1523-536x.1999.00011.x. PMID 10352050
- [Result] Macarthur AJ, Macarthur C. Incidence, severity, and determinants of perineal pain after vaginal delivery: a prospective cohort study. Am J Obstet Gynecol. 2004 Oct;191(4):1199-204. doi: 10.1016/j.ajog.2004.02.064. PMID 15507941
- [Result] Williams A, Herron-Marx S, Carolyn H. The prevalence of enduring postnatal perineal morbidity and its relationship to perineal trauma. Midwifery. 2007 Dec;23(4):392-403. doi: 10.1016/j.midw.2005.12.006. Epub 2006 Dec 29. PMID 17196714
- [Result] Hedayati H, Parsons J, Crowther CA. Rectal analgesia for pain from perineal trauma following childbirth. Cochrane Database Syst Rev. 2003;(3):CD003931. doi: 10.1002/14651858.CD003931. PMID 12917995
- [Result] Chou D, Abalos E, Gyte GM, Gulmezoglu AM. Paracetamol/acetaminophen (single administration) for perineal pain in the early postpartum period. Cochrane Database Syst Rev. 2013 Jan 31;(1):CD008407. doi: 10.1002/14651858.CD008407.pub2. PMID 23440827
- [Result] Gilman G. Drug absorption, bioavailability, and routes of administration. The pharmacological basis of therapeutics. 8th Edition. New York: Macmillan Publishing Co. 1990:7.